CLINICAL TRIAL: NCT06008418
Title: Using Mixed-methods Approach to Explore Health Communication in Hospice Out-Patient Settings (HOUSE): From Middle-range Theory to Clinical Practice
Brief Title: Using Mixed-methods Approach to Explore Health Communication in Hospice Out-Patient Settings
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202303076RINB
Record Dates: First submitted 2023-07-30; First posted 2023-08-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Communication; Palliative Care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Once the patients agree to participate and provide written consent, participants will be assigned to a comparison group or treatment group according to the time of their outpatient appointment. Specifically, during the nine-month period of recruitment, the comparison group participants will be recruited during the first half of the period; and the experimental group will be recruited in the next half of the period. The reason of assigning participants according to time rather than randomization is because of the possible contamination. Because the intervention is designed to be interactive, the intervention will affect not only participating patients' communication behavior but also the physician's behavior.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The LINE Chatbot (Experimental): Participants of the experimental group are required to use the Chatbot before discussing with their physicians.
  Outcome variables are mainly measured at three points: baseline (immediately before the outpatient visit), 24 hours within the outpatient visit, and a week after. At baseline, participants provide their demographic information and complete questionnaires to evaluate their communication self-efficacy and quality of life. After 24 hours, participants are invited to evaluate their satisfaction, communication self-efficacy, shared-decision making process, and the experience of illness invalidation. After a week, the research assistant will remind the participant to evaluate their quality of life. Finally, a retrospective chart review will be conducted one month after the visit to confirm any emergency department visits. Except for the demographic variables (i.e., age, sex, educational level, and diagnosis) and emergency visits.
  Interventions: Behavioral: The LINE Chatbot
- Routine (No Intervention): The comparison group participants will receive routine care (i.e., oral instruction regarding the overall process of outpatient department visits).
  Outcome variables are mainly measured at three points: baseline (immediately before the outpatient visit), 24 hours within the outpatient visit, and a week after. At baseline, participants provide their demographic information and complete questionnaires to evaluate their communication self-efficacy and quality of life. After 24 hours, participants are invited to evaluate their satisfaction, communication self-efficacy, shared-decision making process, and the experience of illness invalidation. After a week, the research assistant will remind the participant to evaluate their quality of life. Finally, a retrospective chart review will be conducted one month after the visit to confirm any emergency department visits. Except for the demographic variables (i.e., age, sex, educational level, and diagnosis) and emergency visits.

INTERVENTIONS:
Behavioral: The LINE Chatbot — The chatbot approach is selected as it uses artificial intelligence to simulate conversations with users. The information can be collected or distributed and even through these conversations trigger human actions. LINE is one of the most widely used freeware applications in Taiwan and its chatbot function is well-organized and relatively easy to modify, adapt, and use. The design of the chatbot aims at the two elements above, ensuring goal alignment and enhancing power sharing, by guiding participants to complete three activities: specifying their goals for today's discussions, providing patient-reported outcomes by self-rating their health-related quality of life, and learning question prompt list based on their needs.
  Arms: The LINE Chatbot

SUMMARY:
This research project aims to investigate health communication in hospice outpatient settings and translate findings into practice by designing and testing a communication aid utilizing health information technology. The specific aims are to: (1) identify the attributes, antecedents, consequences, and implications of the concept of illness invalidation; (2) construct a theoretical framework to describe patient-healthcare provider communication; and (3) based on the theoretical framework, establish a tailored communication aid using health information technology; and investigate its effects on patient outcomes, including (a) satisfaction, (b) communication self-efficacy, (c) illness invalidation, (d) shared-decision making experience, (e) health-related quality of life, and (f) emergency room visits.

DETAILED DESCRIPTION:
While health communication is an established field with numerous publications over decades, it is still hard to conceptualize health communication, including the antecedences and consequences of real communication episodes. Before the mid-1900s, the concept of health communication was more like a "common sense" or was pushed to the background as the focus of medicine was on body systems or cell structure, rather than the whole person. Also, the asymmetric nature of the patient-physician relationship contributes to the ignorance of the quality of health communication. Along with the rise of the idea of "marketing," health communication became a distinct field when hospitals considered patients as consumers since 1960s. Health communication is defined as "a multifaceted and multidisciplinary field of research, theory, and practice concerned with reaching different populations and groups to exchange health-related information…in order to influence, engage, empower, and support individuals, communities, health care professions…" By 1990s, the development and importance of the field of health communication was established as the ideal of patient-centered care has become the norm. The number of relevant research has grown since then and reached a peak in 2018. Interestingly, the amount of published health communication studies has decreased continuously after 2019, despite the constant focus on patient-centered, patient empowerment, and shared-decision making. There is even fewer studies addressed populations with diverse culture background or frontline health communication scenarios. The lack of updated evidence in the field contributes to the fragmental knowledge, including not reflecting the impacts of social and technology changes on health communication and theories that can be easily applied to clinical practice.

The lack of interpersonal communication theories considering real-life medical encounters. As described in the definition of health communication, health communication is a multidisciplinary field which can be observed from its complicated theory background. Theories related to interpersonal health communication were often borrowed from behavioral and social science, medical models, or interpersonal communication filed. These theories can be roughly categorized in to two groups: theories that are more related to interpersonal or mass communication. The two groups were distinguished based on accessibility and message personalization. Because this research project focus on patient-provider communication, the following paragraphs mainly discuss evidence related to interpersonal communication which limits accessibility to a smaller group of people and enable more personalized message.

Except for some theories developed in the interpersonal communication field, most theories that were used to guide health communication research does not address communication directly. For example, health believe model, a theory established in behavioral and social science, has been frequently used to observe the impacts of health communication. Nevertheless, none of the key concepts of health believe model was directly linked to communication. Although communication certainly plays important roles in health beliefs, it is difficult to evaluate or improve real patient-provider communication based on health believe model. Although theories developed by interpersonal communication scholars do address communication goals, process, or outcomes directly, there is still a gap between theory and practice. For example, the majority of these interpersonal communication theories were tested in non-medical encounters. Medical encounters differ than other types of encounters in its therapeutic relationship, unequal power, and special goals and environment. It is hard to apply findings derived from other types of encounters to medical encounters. The remaining few interpersonal theories that specifically address medical encounters, such as uncertainty management theories, action-implicative discourse analysis theory, and multiple goals theory, are probably the most appropriate framework to guide practice and research relevant to real patient-provider communication. However, these theories either only look at special, single concept (e.g., uncertainty in uncertainty management theories, goals in multiple goals theory) or belong to grand theory without describing specific relationships between concepts. There is a scant of literature or framework describe patient-provider communication as a whole, including special concepts and their relationships.

Challenges to patient-provider communication are changing and continue to exist. In the early 21st century, one of the major communication problems between provider and patient is related to physician dominance and physician-centered. While the concept of patient-centered care has been advocated, recent research still indicate that physicians failed to elicit patients' agenda in over half of the medical encounters. Similar to international scholars' findings, previous study also showed questionable communication quality in Taiwan's outpatient settings. Specifically, while patients and caregivers had high level of agreement regarding symptom evaluation, the agreement of symptom evaluation between patients and healthcare providers was not optimal. These challenges support the needs to continuously and intensely examine patient-provider communication theory and practice.

The overall aim of this research project is to investigate health communication in hospice outpatient settings and translate findings into practice by designing and testing a communication aid utilizing health information technology. The specific aims are to: (1) identify the attributes, antecedents, consequences, and implication of the concept of illness invalidation; (2) construct a theoretical framework to describe patient-healthcare provider communication; and (3) based on the theoretical framework, establish a tailored communication aid using health information technology.

ELIGIBILITY:
Inclusion Criteria:

1. terminally ill with a life expectancy of 6 months or less
2. 18-year-old or older
3. able to communicate using Mandarin or Taiwanese

Exclusion Criteria:

* Patients who are not able to use electronic devices due to physical, psychological, or cognitive issues will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Communication self-efficacy(before) | immediately before outpatient visit (T0)
  Before the outpatient visit, communication self-efficacy will be measured by Perceived Efficacy in Patient-Physician Interactions Scales (Chinese version). Knowing the patients' baseline of self-efficacy in "obtaining medical information and attention to their medical concerns from physicians". Ranging from 0 to 10, patients rate from no confidence to extremely confidence to interact with healthcare providers. The total score range between 0 and 100.
Symptoms and quality of life(before) | immediately before outpatient visit (T0)
  Before the outpatient visit, health-related quality of life will be measured by European Organization for Research and Treatment of Cancer (Taiwan Chinese version). Knowing the patients' baseline of functions, symptoms, and overall quality of life. Patients' function and symptom sub-scales are measured by a 4-point Likert scales while overall quality of life sub-scale is measured by a 7-point Likert scales. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.
Subjects satisfaction | 24 hours after the outpatient visit (T1)
  After 24 hours of the outpatient visit and using the LINE chatbot device, satisfaction will be measured by the Chinese Patients' Satisfaction Scale.
  It contains eight aspects (i.e., professionalism, hospitality, patience, efficiency, respect, responsibility, fairness, and ethics) of patients' satisfaction by using a 5-point Likert scale (a higher score means more satisfaction).
Communication self-efficacy(after) | 24 hours after the outpatient visit (T1)
  After 24 hours of the outpatient visit and using the LINE chatbot device, communication self-efficacy will be measured by Perceived Efficacy in Patient-Physician Interactions Scales (Chinese version). Change from the patients' baseline of self-efficacy in "obtaining medical information and attention to their medical concerns from physicians". Ranging from 0 to 10, patients rate from no confidence to extremely confidence to interact with healthcare providers. The total score range between 0 and 100.
Decision making process | 24 hours after the outpatient visit (T1)
  After 24 hours of the outpatient visit and using the LINE chatbot device, the quality of shared-decision making will be measured by the 9-item Shared Decision-Making Questionnaire. Shared-decision making uses a 6-point Likert scale (from completely disagree to completely agree). The total raw score is between 0 and 45 and will be transformed to range from 0 to 100 by multiplying the raw score by 20/9.
Invalidation experience | 24 hours after the outpatient visit (T1)
  After 24 hours of the outpatient visit and using the LINE chatbot device, invalidation experience will be assessed by the Illness Invalidation Inventory. The outcome of patients' perceptions of discounting and lack of understanding will use a 5-point Likert scale questionnaire. Total score range between 8 and 40 with a higher score representing a higher level of invalidation.
Symptoms and quality of life(after) | A week after the outpatient visit (T2)
  After a week of outpatient visit, health-related quality of life as assessed by European Organization for Research and Treatment of Cancer (Taiwan Chinese version). Change from the baseline of patients' functions, symptoms, and overall quality of life. Patients' function and symptom sub-scales are measured by a 4-point Likert scales while overall quality of life sub-scale is measured by a 7-point Likert scales. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.
Provider-patient communication dynamic experience | within 1 year
  A grounded theory approach will be used to construct a theoretical framework for provider-patient communication. The process is fundamental to human experience and advocates developing theories grounded in data. The aim focuses on exploring provider-patient communication, which is a dynamic process.

CONTACTS AND LOCATIONS:
Overall Officials: National Taiwan University Hospital, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan